CLINICAL TRIAL: NCT05817201
Title: A Phase II and III, Randomized, Multicenter Clinical Study: Toripalimab Plus Radiotherapy for Elderly Esophageal Cancer Patients Treated With Non-chemotherapy Strategy
Brief Title: Toripalimab Plus Radiotherapy for Elderly Esophageal Cancer Patients Treated With Non-chemotherapy Strategy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Head of Department of Radiation Oncology, Taizhou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREEN Trial
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Cancer; Radiation Therapy; Immunotherapy; Chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — toripalimab; Tegafur; S 1 (combination); Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab & Radiotherapy (Experimental): Toripalimab, 240mg/d, radiotherapy D7, D28; Thoracic radiotherapy, 54Gy/25F, IMRT; Maintenance Toripalimab therapy after completed radiotherapy, 240mg/Q3W, until progression or 1 years or intolerant
  Interventions: Drug: Toripalimab; Radiation: IMRT
- Chemotherapy & Radiotherapy (Active Comparator): Tegafur, 70mg/m2/d, radiotherapy D1-14, D29-42; Thoracic radiotherapy, 54Gy/25F, IMRT.
  Interventions: Drug: Tegafur; Radiation: IMRT

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg day7 and day 28，every 3 weeks 1month after radiotherapy，until progression or 1 years or intolerant.
  Other Names: JS001; TAB001
  Arms: Toripalimab & Radiotherapy
Drug: Tegafur — Tegafur 70mg/m2/day day 1 to day 14，and day 29 to day42.
  Other Names: S-1
  Arms: Chemotherapy & Radiotherapy
Radiation: IMRT — PGTV 54Gy/2.16Gy/25F/5W, PTV 45Gy/1.8Gy/25F/5W
  Other Names: Irradiation; intensity modulation radiation therapy

SUMMARY:
The goal of this clinical trial is to explore the therapeutic efficacy of immune checkpoint inhibitors combined with radical radiotherapy in elderly patients with esophageal cancer.

DETAILED DESCRIPTION:
Older patients with esophageal cancer are universally intolerant to chemotherapy.

This study is performed to explore a non-chemotherapy strategy for elderly esophageal cancer patients.

Participants will be treated with Toripalimab monoclonal antibody maintenance versus S-1 combined with radiotherapy, intended to explore the efficacy and safety of non-chemotherapy strategy for elderly esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Carcinoma of the esophagus confirmed histologically or cytologically. Lesions that can be measured according to the RECIST standard. AJCC/UICC Staging of Esophageal Carcinoma (Sixth Edition) Clinical Staging Ⅱa to Ⅲ.

Age ≥ 70 years ≤ 85 years old. The ECOG physical state score is 0 to 1. No esophageal perforation, active esophageal bleeding, or significant invasion of trachea or thoracic aorta.

Patients with not previously received chest radiation and speech therapy, immunotherapy, or biological therapy.

Hemoglobin ≥ 100g/L, platelets ≥ 100 * 10^9/L, absolute neutrophil count ≥ 1.5 * 10^9/L。 Serum creatinine ≤ 1.25 times UNL or creatinine clearance ≥ 60 mL/min. Serum bilirubin ≤ 1.5 times UNL, AST (SGOT) and ALT (SGPT) ≤ 2.5 times UNL, and alkaline phosphatase ≤ 5 times UNL.

No history of interstitial pneumonia or previous interstitial pneumonia. FEV1>0.8L。

The patient signs a formal informed consent form.

Exclusion Criteria:

Patients with chest radiation, chemotherapy, or surgical resection of esophageal cancer before the start of this trial Patients with multifocal esophageal cancer, and the lower boundary of the primary lesion of the esophagus is less than 3cm from the esophageal gastric junction.

Patients with severe cardiovascular or pulmonary disease, interstitial pneumonia, or a previous history of interstitial pneumonia.

Patients with obvious esophageal ulcer, moderate or above pain in chest and back, and symptoms of esophageal perforation.

Patients who cannot understand or may not comply with the test requirements. Patients with other malignant lesions, except for curable skin cancer (non melanoma), cervical carcinoma in situ or malignant disease that has been cured for ≥ 5 years.

Researchers believe that some obvious diseases should be excluded from this study.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time Frame: 2 years
  The OS was defined as the duration from the date of of initiation of treatment to the date of death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progression-Free survival | Time Frame: 2 years
  Progression-free survival (PFS) will be calculated from the date of initiation of treatment until the day of documented failure (local recurrence or metastasis occurrence) or until the date of the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Taizhou Enze Medical Center(Group) Enze Hospital Yang, MD, Principal Investigator — Taizhou Enze Medical Center Group
Locations (2):
- China (2):
  - Haihua Yang, Taizhou, Zhejiang
  - Taizhou Enze Medical Center(Group) Enze Hospital, Taizhou, Zhejiang